CLINICAL TRIAL: NCT05014477
Title: Device Embolization After Percutaneous Left Atrial Appendage Occlusion: Risk Factors, Approaches and Outcomes
Brief Title: Therapy Strategies After LAA Occluder Device Embolization
Acronym: LAAODE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cardiovascular Center Frankfurt (Other)
Collaborators: Kerstin Piayda, CardioVascular Center Frankfurt, Frankfurt, Germany (Unknown); Kolja Sievert, CardioVascular Center Frankfurt, Frankfurt, Germany (Unknown); Roberto Galea, Universitätsspital Bern, Bern, Switzerland (Unknown); Moniek Maarse, St. Antonius Ziekenhuis, Nieuwegein, Netherlands (Unknown); Sheba Medical Center (Other Government); Andrey Osadchiy, City Hospital #40, St. Petersburg, Russia (Unknown); Andrey Kalemberg, National Research Center, Moscow, Russia (Unknown); Jung-Sun Kim, Yonsei University Hospital, Seoul, South Korea (Unknown); Aarhus University Hospital (Other); Sajjad A Sabir, Cooper University Hospital, NJ, USA (Unknown); Ashish Pershad, Banner Health, Phoenix, Arizona, USA (Unknown); Markus Sandri, Herzzentrum Leipzig, Leipzig, Germany (Unknown); Jens-Erik Nielsen-Kudsk, University Hospital Aarhus, Aarhus, Denmark (Unknown); George Mark, The Heart House/Cooper University Camden, NJ, USA (Unknown); Dhiraj Gupta, Liverpool Heart and Chest Hospital, Liverpool, UK (Unknown); Pradhum Ram, Emory University, USA (Unknown); Rigshospitalet, Denmark (Other); Norbert Klein, Klinikum St. Georg, Leipzig, Germany (Unknown); Josep Rodes, Laval Hospital, Quebec, Canada (Unknown); Shazia Afzal, Heinrich-Heine University, University Hospital, Duesseldorf (Unknown); Xavier Millán Alvarez, Hospital de la Santa Creu i Sant Pau, Barcelona, Spain (Unknown); James E. Harvey, WellSpan Health, York, PA, USA (Unknown); Wern Yew Ding, University of Liverpool, Liverpool, UK (Unknown); Adel Aminian, Centre hospitalier universitaire de Charleroi, Brussels, Belgium (Unknown); Pamela Moceri, Hopital Pasteur 1, Nice, France (Unknown); Ibrahim Akin, Universitätsmedizin Mannheim, Germany (Unknown); Jacques Mansourati, Hôpital de la Cavale Blanche, Brest, France (Unknown); Eloi Marijon, Hôpital Européen Georges-Pompidou HEGP, Paris, France (Unknown); Ignacio Amat Santos, University Clinical Hospital of Valladolid, Valladolid, Spain (Unknown); Hana Vaknin Assa, Beilinson Hospital, Israel (Unknown); Thomas Robert Schmidt, Herzzentrum Dresden GmbH Universitätsklinik, Dresden, Germany (Unknown); Ran Kornowski, Rabin Medical Center, Petah Tiqwa, Israel (Unknown); Giacomo Boccuzzi, Ospedale san Giovanni Bosco, Torino, Italy (Unknown); Christopher R. Ellis, Vanderbilt University, Nashville, TN, USA (Unknown); Henning Ebelt, Katholisches Krankenhaus St. Nepomuk, Erfurt, Germany (Unknown); Guy's and St Thomas' NHS Foundation Trust (Other); Sonja Lehmann, Hôpital Fribourgeois, Freiburg, Swizerland (Unknown); Oh-Hyun Lee, Yonsai University Hospital, Yongin, Korea (Unknown); Wendy Schell, Cooper University Hospital, NJ, USA (Unknown); Domenico della Rocca, St David's Medical Center, Austin, Texas, USA (Unknown); Pablo Pinon Esteban, Hospital Universitario A Coruña, Spain (Unknown); Jose Gabriel Galache Osuna, Miguel Servet University Hospital, Zaragoza, Spain (Unknown); Enio Guerios, Hospital Pilar, Curitiba, Brazil (Unknown); Nicolas Amabile, Institut Mutualiste Montsouris, Paris, France (Unknown); Ignacio Cruz Gonzalez, University Hospital of Salamanca, Castillay Leon, Spain (Unknown); Weita Chen, Taipei Municipal Wanfang Hospital, Taipei, Taiwan (Unknown); Sandeep Kumar Goyal, Piedmont Heart Institute Buckhead, Atlanta, GA, USA (Unknown); Francesco Gianni, Maria Cecilia Hospital, Cotignola, Italy (Unknown); Máximo Rivero Ayerza, Ziekenhuis Oost Limburg, Genk, Belgium (Unknown); Carsten Skurk, Charité, Universitätsmedizin Berlin, Berlin, Germany (Unknown); Martin Langel, Klinikum St. Georg, Leipzig, Germany (Unknown); Livia Gheorghe, Hospital de la Santa Creu I Santa Pau, Barcelona, Spain (Unknown); Lino Santos, Centro Hospitalar Vila Nova de Gaia, Vila Nova de Gaia, Portugal (Unknown); Royal Victoria Hospital, Belfast (Other); Luis Nombela-Franco, Hospital Clínico San Carlos, Madrid, Spain (Unknown); Francesco Nappi, Centre Cardiologique du Nord de Saint-Denis, Paris, France (Unknown); Matteo Montorfano, Ospedale San Raffaele, Segrate, Milan, Italy (Unknown); Juan Fernández-Armenta, Hospital Universitario Puerta del Mar, Cádiz, Spain (Unknown); Michael Kühne, Universitätsspital Basel, Basel, Swizerland (Unknown); Jesper van der Pals, Lund University Hospital, Lund, Sweden. (Unknown); Can Yücel Karabay, Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Center, Istanbul, Turkey (Unknown); Marco Ancona, San Raffaele Scientific Institute, Milan, Italy (Unknown); Ghassan Moubarak, Clinique Ambroise Paré, Neuilly-sur-Seine, France (Unknown); Tom De Potter, OLV Hospital, Aalst, Belgium (Unknown); Mathieu Lempereur, CHU de Liège, Belgium (Unknown); Clinton Health Access Initiative Inc. (Other); Evgeny Merkulov, Scientific Research Center, Moscow, Russia (Unknown); Liesbeth Rosseel, ASZ Aalst, Belgium (Unknown); Antti Saraste, Heart Center, Turku University Hospital, Turku, Finland (Unknown); Ahmet Güner, Mehmet Akif Ersoy Hospital, Turkey (Unknown); Achille Gaspardone, San Eugenio Hospital ASL Roma, Italy (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Horst Sievert, Principle Investigator, Cardiovascular Center Frankfurt
Other Study IDs: CVC-003
Record Dates: First submitted 2021-08-12; First posted 2021-08-20 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Left Atrial Appendage Occluder; Device Embolisation; Therapy Strategies; Risk Factors
Keywords: left atrial appendage occluder; device embolization; therapy strategy; risk factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients experiencing device embolization after left atrial appendage occlusion: Device embolization following either surgical or interventional left atrial appendage occlusion
  Interventions: Procedure: Removal or leaving of LAA occluders

INTERVENTIONS:
Procedure: Removal or leaving of LAA occluders — After LAA device embolization there are different approaches to dealing with the occluder dislocation. The aim is to find out which way leads to the best outcomes.

SUMMARY:
The investigators thought to evaluate risk factors, therapeutic approaches and outcomes after left atrial appendage occluder device embolization (LAAO, either surgical or interventional).

DETAILED DESCRIPTION:
The global burden of atrial fibrillation (AF) is high, and AF represents a major cause of morbidity, mortality and health-care expenditure. Thromboembolic stroke may be one of the fatal complications and oral anticoagulation has been the mainstay therapy for decades to mitigate stroke risk. However, in poor candidates for long-term anticoagulation (i.e. high bleeding risk, poor drug tolerance or adherence), non- pharmacological stroke prevention with percutaneous left atrial appendage occlusion (LAAO) is a considerable treatment option.

Occluders are implanted into the left atrial appendage (LAA) but they might dislocate and therefore embolize subsequently. In this case, surgical or percutaneous removal of the device may be indicated. Depending on the patient's status, implanting another device can be an alternative to returning to anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients after interventional or surgical left atrial appendage occlusion with device embolization

Exclusion Criteria:

* n/a

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after interventional or surgical left atrial appendage occlusion with device embolization
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedural mortality | In-hospital stay, assessed up to 30 days
  all-cause mortality during the index procedure, any procedure-related death within 30days or during in-hospital stay for the index procedure (if>30days)
Need for cardiac surgery | In-hospital stay, assessed up to 30 days
Catheter-based retrieval of LAA Occluder | up to 5 years (after device implantation)
  peri-procedural device removal

SECONDARY OUTCOMES:
Further complications | up to 5 years (after device implantation)
  Any other complications after device embolization (i.e., thromboembolic events, circulatory problems, CPR etc.)
Risk factors | up to 30 days (after device implantation)
  Favoring conditions for LAAO device dislocation (e.g., anatomical risk factors, risk factors related to the initial procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Eppinger, Principal Investigator — CardioVascular Center (CVC) Frankfurt, Seckbacher Landstraße 65, 60389 Frankfurt am Main, Hesse, Germany
Locations (1):
- CardioVascular Center (CVC) Frankfurt, Frankfurt on the Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided